CLINICAL TRIAL: NCT05903872
Title: EFFECTS OF AROMATHERAPY MASSAGE ON LACTATION IN NON-BREASTFEEDING MOTHERS WITH PREMATURE NEWBORNS IN NEONATAL INTENSIVE CARE UNIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, İlkay Güngör Satılmış, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IGungorSatilmis
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: LACTATION IN MOTHERS WITH PREMATURE NEWBORNS
Keywords: AROMATHERAPY; MASSAGE; LACTATION; BREASTFEEDING
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The sample of the study included a total of 36 postpartum mothers with preterm newborns in 2 groups
  18 mothers in aromatherapy massage group 18 mothers in back massage group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aromatherapy massage group (Experimental): For three days, twice a day (15 minutes each), aromatherapy massage was applied with a mixture of lavender, fennel and frankincense essential oils in almond oil as a carrier oil.
  Interventions: Other: aromatherapy massage
- back massage group (Active Comparator): For three days, twice a day (15 minutes each), back massage was applied using only 1 tablespoon of almond oil (a carrier oil) in order to evaluate the effect of essential oils.
  Interventions: Other: back massage

INTERVENTIONS:
Other: aromatherapy massage — aromatherapy massage was applied using essential oils
  Arms: aromatherapy massage group
Other: back massage — back massage was applied using only almond oil
  Arms: back massage group

SUMMARY:
This study was planned as a randomized controlled experimental study to investigate the effects of aromatherapy massage on lactation in non-breastfeeding mothers with premature newborns in neonatal intensive care unit.

The population of the research, was consisted of all mothers who gave birth preterm in a city hospital in Istanbul between October 2022- April 2023. The sample of the study included a total of 36 mothers (18 in aromatherapy group, 18 in the massage group) who were randomly selected among the mothers who were over 18 years of age, had preterm (<37 weeks) cesarean section, had a single pregnancy, were on the first postpartum day, were asked to express their milk because of the baby's condition, and volunteered to participate in the study.

The data of the study were collected with Participant Characteristics Form, Depression-Anxiety-Stress Scale (DAS-21), Lactation Onset Symptoms Evaluation Form, Milking Follow-Up Form and Visual Analog Scale (VAS) satisfaction evaluation form.

The Participant Characteristics Form and the Depression Anxiety Stress Scale were administered to all mothers within the first 6-8 hours post-operatively, and manual milking training was given. For three days, twice a day (15 minutes each), aromatherapy massage was applied with a mixture of lavender, fennel and frankincense essential oils in almond oil as a carrier oil, while mothers in the massage group were only massaged with almond oil, which is only the carrier oil. Lactation symptoms were evaluated after the massage in both groups and the expressed milk amount was recorded after milking both breasts for at least 15 minutes. In addition, all mothers expressed their milk 8 times a day and recorded the total amount of milk in 24 hours. After the last application, their satisfaction with the application was evaluated with VAS. Descriptive statistical methods, chi-square, Mann Whitney and Friedman tests were used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

* the mothers who were over 18 years of age, had preterm (<37 weeks) cesarean section, had a single pregnancy, were on the first postpartum day, were asked to express their milk because of the baby's condition, and volunteered to participate in the study.

Exclusion Criteria:

* those with breast problems,
* who have allergic reaction to aromatherapy oils,
* using supplements for milk production,
* those who do not like aromatherapy oils or massage
* mothers who do not want to continue tthe study,
* developing postpartum health problems
* and mothers who cannot adapt to manual milking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
the amount of expressed milk | up to 24 hours
  the amount of expressed milk by manual milking

SECONDARY OUTCOMES:
Lactation symptoms evaluated after the massage sessions | twice a day for 3 days
  Lactation symptoms in breasts

OTHER OUTCOMES:
maternal satisfaction survey | at the end of 3rd day
  satisfaction with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Damla Nur Aksaray, MSc, Principal Investigator — Istanbul University-Cerrahpaşa Women Health and Gynecologic Nursing Master Student
Locations (1):
- İstanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No